CLINICAL TRIAL: NCT07063888
Title: A Prospective Phase II Study of Adjuvant Concurrent Chemoradiotherapy With Simultaneous Integrated Boost Following Hepatectomy for Intrahepatic Cholangiocarcinoma With Narrow Margin or Nodal Involvement
Brief Title: A Prospective Phase II Study of Postoperative Concurrent Chemoradiotherapy in Patients With Intrahepatic Cholangiocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, BO CHEN, Associate Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC5322
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Intrahepatic Cholangiocarcinoma (Icc); Adjuvant Chemoradiotherapy; Narrow Margin; Lymph Node Involvement
MeSH Terms: conditions — Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adjuvant Concurrent Chemoradiotherapy with Simultaneous Integrated Boost (Experimental)
  Interventions: Radiation: Adjuvant Concurrent Chemoradiotherapy with Simultaneous Integrated Boost

INTERVENTIONS:
Radiation: Adjuvant Concurrent Chemoradiotherapy with Simultaneous Integrated Boost — Eligibility patients will receive IMRT or VMAT. The prescription dose to high-risk area of tumor bed or positive lymph node was planned at 55-60Gy and the prescription dose to lymphatic drainage regions was planned at 40-45Gy in 20-25 fractions. During radiotherapy, patients will concurrently receive capecitabine (1600 mg/m² on days 1-14, every 21 days for 2 cycles). After radiotherapy, maintenance therapy with capecitabine will continue (2000 mg/m² on days 1-14, every 21 days for 6 cycles). For patients who cannot tolerate capecitabine, S-1 will be used as an alternative.

SUMMARY:
This is a single-arm prospective phase II clinical trial to investigate the efficacy and safety of adjuvant concurrent chemoradiotherapy with simultaneous integrated boost following hepatectomy for intrahepatic cholangiocarcinoma with narrow margin (<1cm) or nodal involvement. Eligibility patients will receive IMRT or VMAT. The prescription dose to high-risk area of tumor bed or positive lymph node was planned at 55-60Gy and the prescription dose to lymphatic drainage regions was planned at 40-45Gy in 20-25 fractions. During radiotherapy, patients will concurrently receive capecitabine (1600 mg/m² on days 1-14, every 21 days for 2 cycles). After radiotherapy, maintenance therapy with capecitabine will continue (2000 mg/m² on days 1-14, every 21 days for 6 cycles). For patients who cannot tolerate capecitabine, S-1 will be used as an alternative. The primary endpoint is 2-year recurrence-free survival. The secondary endpoints are 2-year overall survival, local-regional control rate and incidence of grade 3 or higher adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years, < 80 years
* Patients with primary surgical treatment
* Postoperative pathology confirmed intrahepatic cholangiocarcinoma
* Postoperative pathology showing narrow resection margin (<1cm) or positive lymph nodes
* R0/R1 resection
* Postoperative Child-Pugh score A5-B7
* Patients meeting either of the following conditions must undergo preoperative or pre-radiotherapy PET-CT to exclude distant metastasis or lymph node metastasis beyond the region from the lower esophagus to the aortic bifurcation

  1. Lymph node metastasis accounting for >50% of dissected nodes
  2. Lymph node metastasis involving the paracardial region or below the renal vein level
* Postoperative contrast-enhanced liver MRI to exclude Intrahepatic satellite nodules
* Recovery from surgery with Eastern Cooperative Oncology Group performance status score of 0-2
* Estimated life expectancy >3 months

Exclusion Criteria:

* History of malignancies, except for basal cell skin carcinoma and in situ carcinoma of the cervix
* Had prior abdominal irradiation
* Had prior liver transplantation
* Had serious myocardial disease or renal failure
* Had moderate or severe ascites with obvious symptoms 4 months after surgery
* Duration from surgery ≥ 4 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2028-05-15 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Two-year Disease-free Survival | up to 24 months
  Disease-free survival was calculated from the date of surgical resection to the date of the first recurrence or death

SECONDARY OUTCOMES:
Two-year Overall Survival | up to 24 months
  Overall survival was calculated from the date of surgical resection to the date of death from any cause
Local-Regional Control Rate | up to 24 months
  Patients with stable disease [SD], partial response [PR] or complete response[CR] were recorded as local control.
Incidence of Grade 3 or Higher Adverse Events | up to 24 months
  Adverse events was evaluated during received protocol therapy according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China